CLINICAL TRIAL: NCT04714489
Title: Scientific Title：A Study on the Registration of The Use of Feilike HeJi in Adults
Brief Title: Public Title：A Study on the Registration of The Use of Feilike HeJi in Adults
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: China Academy of Chinese Medical Sciences (Other)
Responsible Party: Principal Investigator, Zhong Wang, Professor, China Academy of Chinese Medical Sciences
Other Study IDs: Felike V1.0
Record Dates: First submitted 2020-12-02; First posted 2021-01-19 (Actual); Last update posted 2021-06-28 (Actual); Status verified 2021-06

CONDITIONS: Bronchial Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Days
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- experimental group
  Interventions: Other: NO.

INTERVENTIONS:
Other: NO. — NO.

SUMMARY:
Feilike HeJi is produced by Guizhou Jianxing Pharmaceutical Co. LTD. For the treatment of phlegm heat caused by lung cough phlegm yellow, bronchial asthma, bronchitis, see the syndrome of proprietary Chinese medicine (approval number: Z20025136) approved by the state and the drug from radix scutellariae, radix peucedani, radix stemonae, red gentian root of deal, phoenix tree, spreading hedyotis herb, red tube 7 flavour, with qingrejiedu, antitussive expectorant effect. In order to fully understand the safety of Feilike HeJi in clinical practice and fulfill the responsibility of production enterprises for patients, the production enterprises initiated this study to further evaluate the safety and understanding of the function characteristics of Feilike HeJi in a wide range of people, so as to guide the clinical rational drug use.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients (age ≥18 years old) who use Feilike HeJi at the specified monitoring time and in the monitoring center (department) ;
* Must voluntarily participate in this study;
* Must meet ethical requirements.

Exclusion Criteria:

* NO

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The users of Feilike HeJi in adults.Patients in this study were sourced from outpatient or/and inpatient wards. Outpatient or inpatient patients are selected according to the Settings of the monitoring points of each research center. In other words, if the monitoring points of a research center are outpatient, the outpatient patients can be registered. If the monitoring site includes outpatient and ward, both outpatient and inpatient will need to be registered. The monitoring points of each research center can be one or more departments.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2021-01-16 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-08-01 (Estimated)

PRIMARY OUTCOMES:
AE | From the prescription of Feilike HeJi to 3 days after stop using Feilike HeJi.
  All the data to be collected are included in Table A and Table B of the registration And Research Information collection of Adults using Feilike HeJi.Data in Table A are filled in by authorized researchers (such as clinicians) and patients, and data in Table B are filled in by authorized researchers (such as clinicians).

CONTACTS AND LOCATIONS:
Overall Officials: Hongchun Zhang, M.D., Study Director — China-Japan Friendship Hospital
Locations (25):
- China (25):
  - China-Japan Friendship Hospital, Beijing, Beijing Municipality
  - Peking University Third Hospital Yanqing Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital Of Guangzhou Medical University, Guangzhou, Guangdong
  - The Eighth Affiliated Hospital, Sun Yat-sen University, Shenzhen, Guangdong
  - Southern University of Science and Technology Hospital, Shenzhen, Guangdong
  - Guizhou Provincial People's Hospital, Guiyang, Guizhou
  - The Second People's Hospital of Guiyang, Guiyang, Guizhou
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - First Affiliated Hospital, Hunan University of Traditional Chinese Medicine, Changsha, Hunan
  - People's Hospital of Ningxiang, Changsha, Hunan
  - Xiangtan County People's Hospital, Changsha, Hunan
  - Nanjing Central Hospital, Nanjing, Jiangsu
  - Yifu Hospital Affiliated to Nanjing Medical University, Nanjing, Jiangsu
  - Nanjing Jiangning Hospital of traditional Chinese Medicine, Nanjing, Jiangsu
  - Guixi People's Hospital, Jiangxi Province, Guixi, Jiangxi
  - Jiangxi University of Traditional Chinese Medicine Affiliated Hospital, Nanchang, Jiangxi
  - Wanzai County People's Hospital, Jiangxi Province, Yichun, Jiangxi
  - Changchun Second Hospital, Changchun, Jilin
  - People's Hospital of Fuxin Mongolian Autonomous County, Fuxin, Liaoning
  - First People's Hospital of Jining City, Jining, Shandong
  - People's Hospital of Mengyin County, Linyi, Shandong
  - Hanyin County People's Hospital, Shaanxi Province, Ankang, Shanxi
  - First Affiliated Hospital of Xi'an Medical College, Xian, Shanxi
  - Peking University Binhai Hospital, Tianjin, Tianjin Municipality
  - Tianjin First Central Hospital, Tianjin, Tianjin Municipality